CLINICAL TRIAL: NCT05574712
Title: An Evolutionary Double Bind Phase II Neoadjuvant Study of Abiraterone Acetate, Leuprolide Acetate, and Belzutifan in Men With Regional Prostate Cancer Eligible for Prostatectomy
Brief Title: A Neoadjuvant Study of Abiraterone Acetate, Leuprolide Acetate, and Belzutifan in Men With Regional Prostate Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Principal Investigator has decided not to activate this trial.
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J2258; IRB00338335 (Other: JHM IRB)
Record Dates: First submitted 2022-10-06; First posted 2022-10-10 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Prostate Cancer
Keywords: prostate; prostate cancer; neoadjuvant; therapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Neoadjuvant Therapy; Leuprolide; Abiraterone Acetate; belzutifan

STUDY DESIGN:
Intervention Model Description: This is an evolutionary double bind, open-label, multi-site, Phase II neoadjuvant study in men with regional prostate cancer planning to undergo prostatectomy. This study will assess the rate of near pathological complete response (pCR) after 3 months (12 weeks) of neoadjuvant treatment with leuprolide acetate, abiraterone acetate, and belzutifan as assessed on prostatectomy specimens.
  Participants will be treated with neoadjuvant therapy for a total of 3 months (12 weeks) prior to prostatectomy. Therapy will consist of leuprolide acetate, abiraterone acetate, and belzutifan. Each drug will be dosed at its respective FDA-approved dose. These dosages are as follows: leuprolide acetate 22.5 mg depot injection x one dose, abiraterone acetate 1000 mg by mouth daily, and belzutifan120 mg administered by mouth once daily. All men will also be treated with prednisone 5 mg by mouth twice daily while on abiraterone acetate in order to blunt its associated mineralocorticoid side effects.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open-Label Treatment Group (Experimental): Participants will be treated with neoadjuvant therapy for a total of 3 months (12 weeks) prior to prostatectomy. Therapy will consist of leuprolide acetate, abiraterone acetate, and belzutifan.
  Interventions: Drug: Neoadjuvant treatment

INTERVENTIONS:
Drug: Neoadjuvant treatment — Each drug will be dosed at its respective FDA-approved dose. These dosages are as follows: leuprolide acetate 22.5 mg depot injection x one dose, abiraterone acetate 1000 mg by mouth daily, and belzutifan120 mg administered by mouth once daily. All men will also be treated with prednisone 5 mg by mouth twice daily while on abiraterone acetate in order to blunt its associated mineralocorticoid side effects
  Other Names: leuprolide acetate; abiraterone acetate; belzutifan

SUMMARY:
For men with prostate cancer that involves the nearby lymph nodes (N1) standard treatment varies. Many men undergo radical prostatectomy (total removal of the prostate) along with the removal of nearby lymph nodes. Other men may opt for androgen deprivation therapy (ADT, a therapy that blocks testosterone) using the two drugs leuprolide and abiraterone - with or without radiation. This research is being done to investigate whether the use of leuprolide and abiraterone, when given in combination with a drug that blocks a molecule that senses oxygen needs by cancer cells, belzutifan, can kill cancer cells in the body prior in men who are planning on having the prostate surgically removed.

DETAILED DESCRIPTION:
Eligible participants will receive 1 dose of leuprolide on day 1 as a subcutaneous injection and abiraterone and belzutifan as pills to take every day for 89 days. Participants will then undergo radical prostatectomy as a standard of care to treat prostate cancer approximately 2 weeks after finishing the study drugs. Participants will have PSA checked 1 year and 2 years after surgery. The list of study procedures (some of which are likely to be part of regular cancer care) will include the collection of data from medical records, imaging tests (CT/MRI/ Prostate-Specific Membrane Antigen Scan PSMA/ Positron Emission Tomography PET CT) to evaluate tumors, and blood collection.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent.
2. Age ≥ 18 years
3. Eastern cooperative group (ECOG) performance status ≤2
4. Documented histologically confirmed adenocarcinoma of the prostate
5. Willing to undergo prostatectomy as primary treatment for localized prostate cancer
6. Regional prostate cancer (per National Comprehensive Cancer Network criteria): T1-4, N1, M0. Patients with negative conventional imaging may have regional prostate cancer defined by PSMA PET imaging.
7. Serum testosterone ≥150 ng/dL
8. Able to swallow the study drugs whole as tablets
9. Willing to take abiraterone acetate on an empty stomach (no food should be consumed at least two hours before and for one hour after dosing).
10. Willing to use a condom if having sex with a pregnant woman, or use a condom and another effective method of birth control if having sex with a woman of childbearing potential. These measures are required during and for one week after treatment with abiraterone acetate.

Exclusion Criteria:

1. Prior local therapy to treat prostate cancer (e.g. radical prostatectomy, radiation therapy, brachytherapy)
2. Prior use of enzalutamide, apalutamide, darolutamide or abiraterone acetate
3. Prior or ongoing systemic therapy for prostate cancer including, but not limited to:

   1. androgen deprivation therapy (e.g. leuprolide, goserelin, triptorelin, degarelix)
   2. Cytochrome CYP-17 inhibitors (e.g. ketoconazole)
   3. Treatment with 1st generation antiandrogen (e.g. bicalutamide) allowed if less than one month of therapy
   4. Immunotherapy (e.g. sipuleucel-T, ipilimumab)
   5. Chemotherapy (e.g. docetaxel, cabazitaxel)
4. Evidence of serious and/or unstable pre-existing medical, psychiatric, or other conditions (including laboratory abnormalities) that could interfere with patient safety or the provision of informed consent to participate in this study.
5. Any psychological, familial, sociological, or geographical condition that could potentially interfere with compliance with the study protocol and follow-up schedule.
6. Abnormal bone marrow function [absolute neutrophil count (ANC)<1500/mm3, platelet count <100,000/mm3, hemoglobin <9 g/dL]
7. Abnormal liver function (bilirubin, Aspartate transaminase (AST), Alanine Transaminase (ALT) ≥ 3 x upper limit of normal)
8. Abnormal kidney function (serum creatinine ≥ 2 x upper limit of normal)
9. Abnormal cardiac function as manifested by the New York Heart Association (NYHA) class III or IV heart failure or history of a prior myocardial infarction (MI) within the last five years before enrollment in the study.
10. History of prior cardiac arrhythmia
11. Baseline pulse oximetry of <90%

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Rate of near pathological complete response (pCR) | 12 weeks
  The rate of near pathological complete response (i.e. ≤5 mm of residual tumor) as assessed on prostatectomy specimens following 3-months (12 weeks) of neoadjuvant leuprolide acetate, abiraterone acetate, and belzutifan.

SECONDARY OUTCOMES:
Negative Margin Rate | 12 weeks
  The negative margin rate as assessed on prostatectomy specimens following 3-months (12 weeks) of neoadjuvant treatment
Rate of Pathologic T3 disease | 12 weeks
  The rate of pathologic T3 disease as assessed on prostatectomy specimens following 3-months (12 weeks) of neoadjuvant treatment.
Rate of radiographic disappearance of prostate nodules | 12 weeks
  Rate of radiographic disappearance of MRI detectable significant prostate nodules (i.e. ≥0.5 cm in size) following 3-months (12 weeks) of neoadjuvant treatment.
Proportion of participants receiving adjuvant radiation therapy | Up to 1 year after prostatectomy
  The proportion of men who receive adjuvant radiation therapy within 1-year of prostatectomy.
Biochemical progression measured by Prostate Specific Antigen (PSA) | 2 years
  The biochemical (i.e. PSA) progression free survival estimate two years after the last patient has accrued (i.e. confirmed PSA post-radical prostatectomy ≥0.2 ng/mL).

OTHER OUTCOMES:
Overall Survival Estimate of Participants | 2 years
  The overall survival estimate two years after the last patient has accrued.

CONTACTS AND LOCATIONS:
Overall Officials: Ken Pienta, M.D, Principal Investigator — Johns Hopkins University